CLINICAL TRIAL: NCT01405898
Title: The Chronic Effects of Beetroot Juice on Circulating Plasma Nitrate and Nitrite Levels and Blood Pressure in Hypertensive Subjects
Brief Title: The Chronic Effects of Beetroot Juice in Hypertensive Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Professor of Vascular Pharmacology, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 08/H0703/91 Chronic
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: hypertension; nitrite; blood pressure; endothelial function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beetroot Juice (Experimental)
  Interventions: Dietary Supplement: beetroot juice
- Nitrate-free beetroot juice (Placebo Comparator)
  Interventions: Dietary Supplement: Nitrate-free beetroot juice

INTERVENTIONS:
Dietary Supplement: beetroot juice — Beetroot juice 4 weeks 250ml daily
  Arms: Beetroot Juice
Dietary Supplement: Nitrate-free beetroot juice — Nitrate-free beetroot juice 4 weeks 250ml daily
  Arms: Nitrate-free beetroot juice

SUMMARY:
We are interested in the effect of diet on blood pressure. Our previous research has shown that beetroot juice lowers blood pressure in healthy people. We now want to see if beetroot juice has this effect in people with high blood pressure. Beetroot juice is naturally rich in nitrate (also found in most other vegetables but particularly in green leafy vegetables). We think that it is the nitrate that lowers the blood pressure.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Healthy adult male and females between 18 and 85 years of age, inclusive.
2. To be eligible, female subjects will be required to state that they are not pregnant, and will not become pregnant during the course of the study.
3. Body mass index (BMI) between 18 and 40 kg/m2
4. A signed and dated written informed consent prior to admission to the study
5. The subject is able to understand and comply with protocol requirements, instructions and protocol---stated restrictions.

and either of the following categories of blood pressure

Category 1---Pre---hypertensive SBP 130---139 or DBP 85---89 on no antihypertensives and will not commence antihypertensives during the course of the study.

Category 2---Grade 1 hypertensive SBP 140---159 or DBP 90---99 on no anti---hypertensives, no target organ damage (TOD), low cardiovascular disease (CVD) risk Category 3---Uncontrolled severe resistant (Grade 3) hypertensive with evidence of difficulty treating to target BP (140/85 or 130/80), with satisfactory adherence to at least one antihypertensive, but insufficient efficacy or intolerance of medications. (Category 3 patients may also be on aspirin and/or a stable dose of cholesterol---lowering medications e.g statins).

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. History of symptomatic coronary artery disease, stroke, or other known atherosclerotic disease.
2. History of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody), or other chronic hepatic disorders.
3. History of increased liver function tests (ALT, AST) due to acute or chronic liver conditions, 3x above the upper limit of normal or bilirubin 1.5x above the upper limit of normal at screening.
4. Renal impairment with creatinine clearance (eGFR) of <50 ml/min at screening.
5. Current poorly controlled diabetes mellitus, defined as HbA1c >10% at Screen.
6. Subjects with LDLc, >7.5 mmol/l. Fasting TG level >6mmol/l.
7. History of heart failure defined as NYHA class II --- IV or those with known severe LV dysfunction (EF<30%) regardless of symptomatic status
8. History of malignancy within the past 5 years, other than non---melanoma skin cancer.
9. Current life---threatening condition other than vascular disease (e.g., very severe chronic airways disease, HIV positive, life---threatening arrhythmias) that may prevent a subject from completing the study.
10. Alcohol or drug abuse within the past 6 months.
11. Use of an investigational device or investigational drug within 30 days or 5 half---lives (whichever is the longer) preceding the first dose of study medication.
12. Subjects who will commence or who are likely to commence treatment with non---steroidal anti--- inflammatory drugs (NSAIDs) (other than aspirin), from screening until study completion.
13. Any non---stable dosing of ongoing medication regimens throughout the study trial.
14. The subject has a three---month prior history of regular alcohol consumption exceeding an average weekly intake of > 28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a half---pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine; or a positive alcohol breath test at the screening visit
15. A positive urine test for drugs of abuse (not related to known medications the subject is taking, i.e., codeine for pain management) or alcohol at screening or prior to study medication administration.
16. Any other subject whom the Investigator deems unsuitable for the study (e.g., due to either medical reasons, laboratory abnormalities, expected study medication noncompliance, or subject's unwillingness to comply with all study---related study procedures).
17. Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
18. Subjects with any acute infection, or significant trauma (burns, fractures).
19. Subjects who have donated more than 500 mL of blood within 56 days prior to the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, Principal Investigator — Queen Mary University London
Locations (1):
- Queen Mary University London, London, London, United Kingdom

REFERENCES:
- [Derived] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976

RESULTS

PARTICIPANT FLOW:
Groups:
- Beetroot Juice: Beetroot juice, 4 weeks 250ml daily
- Nitrate-free Beetroot Juice: Nitrate-free beetroot juice, 4 weeks 250ml daily
Period: Overall Study
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Started | 34 | 34
Completed | 32 | 32
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (13.9) | 56.3 (16.4) | 56.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Difference in Change in Clinic Systolic Blood Pressure From Baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
mmHg | -8.7 (8.2) | -1.0 (8.4)

2. Secondary Outcome: Difference in Change in Plasma Nitrite Concentration From Baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
umol/L | 0.53 (0.37) | 0.01 (0.16)

3. Secondary Outcome: Difference in Change in Endothelial Function From Baseline
Description: as measured by flow-mediated dilatation [%change in diameter of vessel] - an increase in diameter demonstrates an improvement in endothelial function
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: % dilatation
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
% dilatation | 0.9 (1.3) | 0.1 (0.6)

4. Primary Outcome: Difference in Change in Clinic Diastolic Blood Pressure From Baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
mmHg | -3.2 (5.4) | -0.7 (4.2)

5. Primary Outcome: Difference in Change in Ambulatory Systolic Blood Pressure From Baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
mmHg | -6.6 (6.5) | 0.8 (4.9)

6. Primary Outcome: Difference in Change in Ambulatory Diastolic Blood Pressure From Baseline
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
mmHg | -4.3 (6.0) | 0.9 (3.8)

7. Secondary Outcome: Difference in Change in Arterial Stiffness From Baseline
Description: carotid-femoral pulse wave velocity [m/s] measured by Vicorder
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Number analyzed (Participants) | 32 | 32
m/s | -0.59 (0.93) | 0.01 (1.11)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Beetroot Juice | Nitrate-free Beetroot Juice
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes